CLINICAL TRIAL: NCT04229719
Title: Effect of Topical Melatonin Application on Dental Implant Osseointegration and Marginal Bone Level (Clinical and Radiographic Evaluation)
Brief Title: Effect of Topical Melatonin Application on Dental Implant Osseointegration and Marginal Bone Level
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Zaid Mohannad Yasser, Bachelor of Dental Surgery (master's student), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U0004TGZ
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Third professional person apply melatonin powder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin group (Experimental): Melatonin powder (N-Acetyl-5-methoxytryptamine) 1.2mg topical application in osteotomy site.
  Interventions: Drug: N-acetyl-5-methoxytryptamine
- Control group (No Intervention): No drug intervention

INTERVENTIONS:
Drug: N-acetyl-5-methoxytryptamine — 1.2 mg of melatonin powder will place in the osteotomy site before the insertion of the implant.
  Other Names: Melatonin powder
  Arms: Melatonin group

SUMMARY:
Background: Melatonin (N-acetyl-5-methoxy-tryptamine) is an indoleamine synthesized and secreted by the pineal gland and other organs, such as the retina, bone marrow, and intestines in a circadian pattern. Some authors claimed that Melatonin induces bone formation, increase bone density, and bone implant contact. According to animal and human studies the melatonin can be used topically during implant placement to increase bone implant contact and reduce marginal bone loss.

Purpose: The aim of this study was to evaluate the effect of the topical administration of melatonin on osseointegration of dental implants and in minimize marginal bone loss.

Materials and Methods: Twenty single-piece endosseous implants (Dentium Co, Korea) will use to restore missing lower teeth from canine to first molar area. The study will be split-mouth technique, each patient serve as his own control (served into 2 groups), the study side (topical application of melatonin in the implant side), and the control side (no melatonin in the other implant side of the same patients).The primary and secondary stability of dental implant will be evaluated by periotest M device and measure bone level as baseline immediately after implant placement and after 6 months follow up by CBCT.

DETAILED DESCRIPTION:
Melatonin (N-acetyl-5-methoxy-tryptamine) is an indoleamine synthesized and secreted by the pineal gland and other organs, such as the retina, bone marrow, and intestines in a circadian pattern. Extrapineal sites contribute poorly, or only upon specific stimuli to circulating melatonin. Melatonin influences numerous physiological actions that may be mediated by the binding of the indoleamine to membrane receptors in all tissues. Because of its lipophilic properties, melatonin passes through cell membranes to gain access to subcellular organelles, being capable to bind to some cytosolic proteins like kinase-C . Currently, melatonin is not considered a hormone in the classical sense of the term, because it is synthesized in several organs and does not exert effects on a specific target , but it is rather a powerful cell protector against molecular damage. For the synthesis of melatonin, the pineal cells take up tryptophan from the blood and, through hydroxylation and a decarboxylation process, turn it into serotonin. Serotonin is then converted into N-acetylserotonin through N-acetyltransferase and subsequently methylated to the final form of melatonin by the enzyme hydroxy indole-O-methyltransferase . In healthy individuals, the maximum secretion of melatonin occurs between midnight and 2 a.m., then it decreases to a minimum during the day. Melatonin has numerous physiological functions in different parts of the body, such as the control of circadian rhythms \, regulation of body temperature, and activation of the immune system.In the oral cavity, melatonin has been recognized as an important substance with paracrine effects on nearby cells, it also acts as an antioxidant and an anti-inflammatory and plays an important role in bone formation and in the reduction of bone resorption.

Osseointegration defined as a direct connection between living bone tissues and a titanium implant without any connective tissues. Osteoblasts are bone formative cells, and osteoclasts are bone resorptive cells. When these cells work together physiologically, the formation and resorption processes of bone tissue is known as bone remodelling. The remodeling of bone tissues is regulated by the action of systemic hormones (estradiol, parathyroid, growth, and melatonin) and by the bone marrow and osteoid matrix-derived growth factors.Insufficient bone quality and quantity can be seen frequently in elderly populations with atrophic and osteoporotic bones, and this situation stems from increased osteoclastic activity due to a reduction in osteoblastogenesis. In addition, local free radical concentrations in all body cells, including osteoblasts, can reduce osteoblastic activity in aged patients. This process could lead to a reduction in bone regeneration capacity. Melatonin can also suppress osteoclastogenesis, and therefore inhibit bone tissue resorption. In addition to this, in vitro research has reported that melatonin can increase osteoblast proliferation and differentiation. So was proposed that the local application of melatonin during surgical implant placement procedures would be an effective treatment technique for dental implant osseointegration. Worthy osseointegration is a prerequisite for dental implants. Optimal osseointegration depends on the formation of new bone around implants, which may be stimulated by the application of biomimetic agents. Considering the bone metabolism, melatonin acts directly on the osteoclast, a multinucleated cell, which resorbs the extracellular matrix through various mechanisms, including the production of free radicals. Moreover, in pre-osteoblast cultures from rats, melatonin, in a dose-dependent manner, promoted the development of bone sialoprotein and other protein bone markers, including alkaline phosphatase, osteopontin, and osteocalcin, and speeds up their period of differentiation into osteoblasts from the normal rate, which is 21 days, to 12 days, this reaction is mediated by the membrane receptors for the indole. Also, melatonin, may interfere with the function of the osteoclast and thereby inhibit bone resorption. conducted an experimental study using melatonin with dental implants in dogs. Two weeks after implant insertion, melatonin significantly increased all parameters of osteointegration. It has been observed that melatonin, increases bone mass by suppressing resorption through down-regulation of the RANKL-mediated osteoclast formation and activation. These data point towards an osteogenic effect of melatonin that may be of clinical importance, as it could be used as a therapeutic agent in situations in which bone formation would be advantageous, such as in the treatment of fractures or of osteoporosis.

Toxicology of Melatonin:- The physiological functions of the pineal hormone melatonin are extremely diverse. The functions include direct and indirect modulations of anti-oxidative defense, blood pressure, body temperature, cortisol rhythm, reproduction and immune function . Correspondingly, exogenous melatonin has been investigated as a treatment for a number of medical and surgical diseases, demonstrating encouraging results . In the USA, melatonin is available as an over-the-counter non-prescription drug. In most European countries, however, melatonin remains a prescription drug (Circadin) and has only been approved as a treatment for primary insomnia in people over 55 years of age. However, a recent Norwegian register study documented a 3- to 5-times increase in off-label use among children and adolescents in the time period 2004 to 2012 . Melatonin is generally considered safe, but the increasing clinical use with potentially increasing doses necessitates further investigations of the risks of both mild and serious adverse effects.

Periotest M device:-

Periotest device was developed to measure the damping characteristics of natural teeth and has been used to evaluate implant. It was developed by Schulte in 1983 to quantify TM , and then utilized by Teerlinck et al , to measure implant stability and to overcome destructive methods in measuring the implant stability like histologic analysis, tensional test, push-out/pull-out test and removal torque analysis. The (Classic/Wired) Periotest device has been the subject of several studies with generally favorable results. These results showed that the Periotest device generally demonstrated a high degree of repeatability and reliability. A wireless version of the Periotest (Periotest "M") has been introduced to the profession. According to information provided by the electronic page of the Periotest M /wireless device manufacturer (Medizintechnik Gulden, Modautal, Germany), Periotest M is simpler to perform an objective evaluation of an implant's stability compared to classic Periotest. In Periotest M wireless design, the user can benefit from maximum freedom of movement. The device can be used for taking measurements on a wide variety of implants, without the need for any special accessories, such as a smart peg . The Periotest has an important advantage against the others like the Osstell device: it can be applied directly to the implant superstructure .

The limitations of Periotest are the inability of the instrument to measure the mesiodistal mobility, the possible effect of position and angle of the rods on the measured value . The readings of PTV are from (-8 to +50) according to information provided by the device manufacturer (Medizintechnik Gulden, Modautal, Germany) .

Cone-beam computed tomography (CBCT):-

Cone-beam computed tomography (CBCT) is an imaging modality that offers significant advantages for the evaluation of implant patients . The field of view (FOV) is an important feature that describes the extent of the imaged volume from large FOV (greater than 15 cm) to medium FOV (8 to 15 cm) and limited FOV (less than 8 cm). Limited FOV units image a small area, delivering less radiation and producing a higher-resolution image . CBCT allows for defining with elevated accuracy the quality (cortical/medullar ratio) and the quantity (height and thickness) of bone available for the implant, providing the essential information of performing or not a preimplant bony graft . when compared to medical CT, CBCT can be recommended as a dose reducing technique for dental implant applications. The effective dose from CBCT examinations ranges from 13 µ Sv with the 3D Accuitomo CBCT machine using the 4 x4 cm FOV to 479 µ Sv with the CB Mercury CBCT machine . For comparison, the effective dose from one panoramic radiograph is approximately 10 to 14µSv. Furthermore, the exposure from a maxillomandibular medical CT ranges from 474 to 1160 µSv. The average background radiation in the United States is 3000 µSv (3 mSv) per year or 8 µSv per day . It is important to understand that every effort must be made to reduce the effective radiation dose to the patient. By using the smallest possible FOV, the lowest mA setting, the shortest exposure time, and a pulsed exposure mode of acquisition, it is possible to accomplish effective dose reduction to the patient.

Twenty single-piece endosseous implants (Dentium Co, Korea) will use to restore missing teeth in the upper or lower jaw (canine to 1st molars area) from both sides. The study will be split-mouth technique, each patient serves as his own control (served into 2 groups), the study side (topical application of melatonin in the implant side), and the control side (no melatonin in the other implant side of the same patients). According to the study reported by (Cutando et al., 2008) the estimated dose of melatonin required to enhance osseointegration of dental implant and minimize the marginal bone resorption is 1.2 mg of melatonin powder for each implant. CBCT for all patients before implant placement to determine bone density, dimension, and anatomical landmarks. Prior to surgery, all patients will instruct to use chlorhexidine 0.12% mouthwash as antiseptic. After local anesthesia, a mucoperiosteal flap will reflect. The manufacturer's instructions should be followed for the preparation of the implant osteotomy site. For the study side, 1.2 mg of melatonin powder will place in the osteotomy site before the insertion of the implant. For the control side, no melatonin powder will be used and implants will be inserted directly in the prepared implant site. After dental implant installation, the gingival former will insert into the body of the fixture, then the Periotest M device will use to measure the primary stability of the DI fixture. After that, the gingival former will be removed and cover screw place and tightened into the fixture. Sutures will place after flap replacement. Patients should be instructed to use antibiotics amoxicillin 500mg and metronidazole 500mg 3 times/day for 5 days after surgical procedure, soft diet and proper oral hygiene measures. Also, CBCT immediately after implant placement to record baseline bone level, CBCT after 6 months follow up to measure marginal bone level around implant comparing with baseline measurement, and measure the secondary stability using periotest M device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have good oral hygiene.
2. Patients were periodontally healthy.
3. Patients had at least two missing teeth in the upper or lower jaw (canine to 1st molar area) indicated for the dental implant.

Exclusion Criteria:

1. Patients with any systemic diseases that influence bone healing such as osteoporosis and diabetes mellitus.
2. Fully edentulous.
3. Patients who had parafunctional habits.
4. Smokers.
5. Patients who were not able to follow the treatment protocol.

   -

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Measuring marginal bone level | 6 months .
  measure crestal bone loss around dental implant using a cone-beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Measuring primary stability of the dental implant | 0 day.
  using periotest M device for measurement.
Measuring secondary stability of the dental implant | 6 months.
  using periotest M device for measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry / University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT04229719/Prot_000.pdf